CLINICAL TRIAL: NCT05762341
Title: Istanbul University Cerrahpaşa Graduate Education Institute, PhD Student
Brief Title: Pressure Injury Training With a Blended Approach Learning Approach on Care Behaviors of Intensive Care Nurses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Ebru Kiraner, specialist nurse, PHD STUDENT, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: IUC Gradu Educ Inst
Record Dates: First submitted 2023-02-28; First posted 2023-03-09 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Pressure Injury
Keywords: "pressure injury", "intensive care nurse" , "prevention"
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Intervention Model Description: Number of groups 2 (experiment, control), number of measurements 2 (pretest, posttest),
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXPERIMENT GROUP (Experimental): BOTH GROUPS WILL RECEIVE PRESSURE INJURY PREVENTION TRAINING. ONLY EXPERIMENTAL GROUP WILL USE THE MOBILE LEARNING TOOL
  Interventions: Other: PRESSURE INJURY PREVENTION TRAINING
- CONTROL GROUP (Experimental): BOTH GROUPS WILL RECEIVE PRESSURE INJURY PREVENTION TRAINING. ONLY EXPERIMENTAL GROUP WILL USE THE MOBILE LEARNING TOOL
  Interventions: Other: PRESSURE INJURY PREVENTION TRAINING

INTERVENTIONS:
Other: PRESSURE INJURY PREVENTION TRAINING — PREVENTION OF PRESSURE INJURY TO FACE TO FACE TRAINING

SUMMARY:
By saving life or delaying death, the length of stay of the patient in the intensive care unit is prolonged, and this leads to the emergence of other problems in addition to the disease in the patient. Pressure injuries are one of these problems. Although many internationally accepted pressure injury prevention guidelines are available, it is frequently reported that there is no significant reduction in pressure injury prevalence. It has been emphasized in the literature that nurses do not have enough knowledge about the prevention of pressure injury. "Blended Learning", in which technologies such as web-based, e-learning and m-learning are used together with face-to-face education, is an effective approach in realizing learning outcomes. This approach facilitates the achievement of the educational program's objectives by integrating the positive aspects of web-assisted learning and face-to-face learning. In the light of these explanations, it is aimed to examine the effect of pressure injury prevention training given with the blended learning approach on the care behaviors of intensive care nurses.

DETAILED DESCRIPTION:
The research was planned in a mixed design with a qualitative dimension in terms of determining the experimental and training needs, using the focus group interview method in the evaluation of the program, with the aim of examining the effect of pressure injury prevention training given with the blended learning approach on the care behaviors of intensive care nurses.The universe of the study consists of a total of 100 nurses working in the 3rd Level intensive care units of Istanbul University-Cerrahpaşa Cerrahpaşa Faculty of Medicine. The sample size of the study was calculated by using power analysis. Since the differences between the experimental and control groups before and after the experiment were examined comparatively in the research, ANOVA will be made for mixed measurements. Accordingly, the sample size was calculated by keeping the effect size (Cohen's f) 0.25, that is, at a medium level, based on the expected averages and standard deviations of the groups. G*Power 3.1.9.4 software (Faul, Erdfelder, Lang & Buchner, 2007) was used for the calculation. In order to make a decision with 95% confidence for Type I, the expected power of α error was 0.05 and for Type II error 1-β expected power was 0.80. When the number of groups was entered as 2 (experiment, control), the number of measurements was 2 (pretest, posttest), the expected correlation between repeated measurements was 0.5, and the ε correction was 1, the expected total sample size for this study was calculated as 34 people. Accordingly, there will be a total of 44 people in the research, 17 people in the experimental and control groups, taking into account the possibility of data loss. In order to prevent interaction between the groups in the formation of the experimental and control groups, it will be randomly assigned by paying attention to the fact that the experimental group is from one unit and the control group is from the other unit. Homogenization will be achieved between the groups in terms of having an intensive care nursing certificate, age, years of experience, years of working in intensive care, and Knowledge Evaluation Scale score in Preventing Pressure Ulcers. It will be collected by the researcher and the nurse in charge of the unit by using the Nurse Information Form, the Information Evaluation Scale in Pressure Ulcer Prevention, the Pressure Injury Prevention Efficiency Evaluation Form, the Training Program Evaluation Form, the Semi-Structured Interview Form before the Training Program, and the Semi-Structured Interview Form after the Training Program.

ELIGIBILITY:
Inclusion Criteria:

* Adult intensive care nurses working in the Third Level intensive care unit,
* have not received pressure injury training in the last year,
* voluntarily agree to participate in the study will be included.

Exclusion Criteria:

* Nurses who received pressure injury training in the last year
* work in the pediatric intensive care unit and neonatal intensive care unit

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-03-14 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
INCREASE IN PRESSURE INJURY PREVENTION BEHAVIOR SCORES | 3 MONTHS LATER
  INCREASED BEHAVIOR SCORES TO BE TAKEN FROM THE PRESSURE INJURY PREVENTION QUALIFICATION FORM

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul university Cerrahpaşa hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No